CLINICAL TRIAL: NCT03324425
Title: A Phase II Single Arm Trial of Adding Simvastatin to Dual Anti-HER2 Therapy in Patients With HER2-Positive Metastatic Breast Cancer
Brief Title: Simvastatin Plus Dual Anti-HER2 Therapy for Metastatic Breast Cancer
Acronym: SIMPHONY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Breast Care Center (Other)
Responsible Party: Principal Investigator, Mothaffar Rimawi, Associate Professor, Baylor Breast Care Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-41818
Record Dates: First submitted 2017-09-26; First posted 2017-10-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Stage IV
Keywords: breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Simvastatin (Experimental): Simvastatin 80 mg in combination with anti-HER2 therapy regimen
  Interventions: Drug: Simvastatin 80mg

INTERVENTIONS:
Drug: Simvastatin 80mg — Participants will receive simvastatin 80 mg by mouth daily at bedtime
  Other Names: Zocor

SUMMARY:
This study recruits patients with metastatic breast cancer who have progressed on their current regimen of dual anti-HER2 therapy. This study evaluates whether or not the addition of simvastatin to the dual anti-HER2 therapy regimen helps make the tumor respond to the anti-HER2 therapy again. All participants will receive simvastatin in combination with their current anti-HER2 therapy regimen.

DETAILED DESCRIPTION:
This study is recruiting participants with metastatic breast cancer that is HER2 positive. "Metastatic" means that cancer has spread to areas of the body outside of the breast. "HER2 positive" means that a cancer cell has too many HER2 receptors on its surface. HER2 receptors act like copy machines, and help tell cancer cells to grow and multiply.

Drugs known as HER2-targeted therapies are often used to treat HER2-positive cancers. HER2-targeted therapies work by blocking the HER2 protein from telling the cell to grow and divide. Once the protein stops working, the cancer cells can no longer make copies of themselves. Once a cancer cell becomes unable to make copies of itself, the tumor will start to shrink. However, some tumors are able to find other ways to make copies of themselves, even when the HER2 protein is blocked. When this happens, the cancer will start to grow again. Researchers believe that adding a drug called simvastatin to an anti-HER2 therapy regimen may cause the cancer to start responding again to your HER2-medications.

Simvastatin is a drug that is approved by the Food and Drug Administration (FDA) to treat high cholesterol. Laboratory research has shown that simvastatin together with dual HER2-targeted therapy slows the growth of breast cancer tumors that had been growing on dual HER2-targeting therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Patients must have histologically confirmed and documented adenocarcinoma of the breast with metastatic disease not amenable to curative therapy.
* Cancer must be HER2-positive, according to ASCO-CAP guidelines. Any ER and PR status is allowed.
* Participants must have documented disease progression while receiving dual anti-HER2 targeted therapy for metastatic breast cancer, as per investigator assessment. Any combination of biologic therapies is acceptable. Prior chemotherapy is acceptable, but patients must have been off cytotoxic chemotherapy for at least 1 month. Patients with ER-/HER2+ disease have must be failed at least 1 line of chemotherapy in the metastatic setting. Patients with ER+/HER2+ disease who progressed on dual anti-HER2 therapy plus endocrine therapy are eligible. Concomitant endocrine therapy is acceptable and may be continued at the discretion of the treating physician.
* Patient must be female and at least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2
* Patients must have measurable disease, per RECIST criteria v1.1.21
* Participants must not have undergone major surgery or radiation therapy within 28 days prior to beginning treatment with simvastatin. Any toxicity from prior surgical or radiation treatment must have sufficiently resolved prior to study entry, as determined by the treating physician.
* Estimated life expectancy of ≥ 12 weeks.
* Ability to swallow oral medications.
* Participants must have adequate organ function as defined by:

  1. ANC ≥1.5 x 109/L, platelet count ≥100 x 109/L, haemoglobin ≥ 10 g/dL.
  2. creatinine < 1.5 x UNL (upper normal limit)
  3. Total bilirubin < 1.5x UNL
  4. ALT & AST < 2.5xUNL; alkaline phosphatase < 2.5xUNL;
  5. Creatine phosphokinase (CPK) ≤ 2.5 x UNL
* Baseline left ventricular ejection fraction (LVEF) ≥ 50% as determined by either echocardiography (ECHO) or multi gated acquisition (MUGA) scan.
* Patients with CNS metastatic disease are allowed if the disease is controlled and stable for at least 3 months by CT or MRI.
* Negative pregnancy test within 7 days prior to study treatment start, for women of childbearing potential. Women of childbearing potential must agree to use an adequate form of contraception for the duration of their study participation

Exclusion Criteria:

* Patients currently treated with a statin or who have been treated with a statin in the past 2 months are ineligible for this study.
* Known hypersensitivity to statins.
* Prior history of rhabdomyolysis.
* Patients who consume more than 3 alcoholic beverages per day.
* Lack of physical integrity of the upper gastrointestinal tract, clinically significant malabsorption syndrome, or inability to take oral medications.
* Poorly controlled hypertension at the physician's discretion or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident (CVA) / stroke within ≤ 6 months prior to the first study treatment, myocardial infarction within ≤ 6 months prior to the first study treatment, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia requiring medication.
* Current severe, uncontrolled systemic disease (e.g. pulmonary, or metabolic disease; wound healing disorders; ulcers; or bone fractures)
* Current or past infection with Human Immunodeficiency Virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
* Receipt of IV antibiotics for infection within 7 days of study enrollment.
* History of other malignancies within the last 2 years, except for carcinoma in situ of the cervix or basal cell carcinoma
* Participants with bone-only disease are excluded, unless a measureable lesion is present, as defined by RECIST 1.1.
* Patients who suffer from a medical or psychiatric condition that, in the opinion of the principal investigator, would impair their ability to participate in the study.
* Concurrent interventional studies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response | Up to approximately 24 months
  Objective response is defined as complete response or partial response, according to RECIST criteria.

SECONDARY OUTCOMES:
Clinical benefit | Up to approximately 24 months
  Clinical benefit is defined as the number of objective responses plus the number of participants with stable disease lasting greater than 24 weeks
Duration of Response | Up to approximately 24 months
  The length of time participants have a partial response, complete response or stable disease prior to disease progression
Time to Progression | Up to approximately 24 months
  The length of time from the start of treatment until the disease starts to get worse or spread to other parts of the body
Number of treatment-related adverse events, as assessed by the National Cancer Institute Common Terminology Criteria v. 4.0 (CTCAE v. 4.0). | Up to approximately 24 months
  This is the number of side effects reported by participants receiving simvastatin in combination with HER2-therapy.
HMG-CoA Reductase and HMG-CoA Synthase 1 protein levels in baseline and post-treatment tumor biopsies | Up to approximately 24 months
  This measures the levels of certain enzymes in a tumor that help scientists understand how simvastatin is affecting the cancer cells.

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Harris Health System - Smith Clinic, Houston, Texas
  - O'Quinn Medical Tower - McNair Campus; Dan L Duncan Comprehensive Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No